CLINICAL TRIAL: NCT02035865
Title: Nevropsykiatri og Hjertetransplantasjon
Brief Title: Mood and Cognitive Outcome After Heart Transplantation (the MOODHEART Study)
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ira Hebold Haraldsen, MD, dr.philos., Oslo University Hospital
Other Study IDs: REK sør-øst 2013/1260
Record Dates: First submitted 2013-12-02; First posted 2014-01-14 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Psychiatric Diagnosis; Cognition Disorders
Keywords: Psychiatric morbidity; Cognitive function; Heart transplantation; Mortality; Cardiac allograft vasculopathy
MeSH Terms: conditions — Mental Disorders; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants from former study 1: Surviving participants from a former study called 'Psykosomale faktorer hos pasienter med hjertesvikt og hos hjertetransplanterte'
- Participants from former study 2: Surviving participants, included at the Norwegian centre, from a study called 'Scandinavian Heart Transplant Everolimus De Novo Study with Early Calcineurin Inhibitor Avoidance (SCHEDULE)' (NCT01266148)

SUMMARY:
The investigators aim at characterizing neuropsychiatric consequences of heart transplantation (HTX) and at assessing the impact of depressive symptoms after HTX on mortality and cardiac allograft vasculopathy (CAV).

ELIGIBILITY:
Inclusion Criteria:

* Participant in one of two former studies and heart transplanted at the time of inclusion into this former study

Exclusion Criteria:

* Cognitively not capable to consent to participation and/or
* Insufficient fluent in the Norwegian language to complete both psychiatric and neuropsychological assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surviving participants from two former studies
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Psychiatric morbidity | At time of enrollment
  Psychiatric diagnoses by clinician and self-rapport
Cognitive function | At time of enrollment
  Neuropsychological assessment

SECONDARY OUTCOMES:
All cause mortality | 14 and 3 years respectively
  Time since enrollment in former study; i.e. approximately 14 years (study 1) and approximately 3 years (study 2)
Cardiac allograft vasculopathy | 14 and 3 years respectively
  Time since enrollment in former study; i.e. approximately 14 years (study 1) and approximately 3 years (study 2)

OTHER OUTCOMES:
Cerebral pathology | At time of enrollment
  MRI of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Ira R. Hebold Haraldsen, MD/dr philos, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway